CLINICAL TRIAL: NCT04072705
Title: A Multicenter Prospective observationaL Study to evAluate the effecT of Clopidogrel on the prEvention of Major vascuLar Events According to the gEnotype of Cytochrome P450 2C19 in Ischemic Stroke paTients; PLATELET Study
Brief Title: Clopidogrel Preventive Effect Based on CYP2C19 Genotype in Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Collaborators: SAMJIN PHARM (Unknown)
Responsible Party: Principal Investigator, Kyung-Yul Lee, KyungYul Lee, Professor, Gangnam Severance Hospital
Other Study IDs: 3-2019-0195
Record Dates: First submitted 2019-08-25; First posted 2019-08-28 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Acute Ischemic Stroke
Keywords: Pharmacogenetics; Cytochrome P450 2C19; Clopidogrel; Stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cytochrome P450 2C19 genotype
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1. Poor and intermediate metabolizer group: Poor and intermediate metabolizer group: acute ischemic stroke patients with poor and intermediate metabolizer genotype of cytochrome P450 2C19 for clopidogrel.
  Interventions: Drug: General principles of care and judgement of researcher
- 2. Extensive metabolizer group: Extensive metabolizer group: acute ischemic stroke patients with Extensive metabolizer genotype of cytochrome P450 2C19 for clopidogrel.
  Interventions: Drug: General principles of care and judgement of researcher

INTERVENTIONS:
Drug: General principles of care and judgement of researcher — Because our study will be performed by observational design, there will be no intervention for our study. Because it is a registry-based study, overall decision making for medications will be performed according to the general principles of care and judgement of researcher.

SUMMARY:
The hypothesis of this study is that "the poor metabolizer or intermediate metabolizer of the cytochrome P450 2C19 genotype in patients with acute ischemic stroke is associated with increased risk of composite cardiovascular events (recurrent stroke, myocardial infarction, cardiovascular death) compared to those who of extensive metabolizer of the cytochrome P450 2C19 genotype".

DETAILED DESCRIPTION:
Clopidogrel, one of the antiplatelet agents used for secondary prevention in patients with ischemic stroke and coronary artery disease, has been shown to have a superior antiplatelet effect compared to aspirin, and is therefore being administered to many patients with stroke and coronary artery disease. Clopidogrel inhibits platelet-derived ADP receptor, P2Y12, in the liver to produce an anti-platelet effect. It has been suggested that clopidogrel resistance could be occurred from drug-drug interaction via the same pharmacological metabolic pathway. Previous studies reported that the genotypes of Cytochrome P450 2C19, which is involved in the metabolism of clopidogrel in the liver, lead to differences in drug response and recurrence rates of cardiovascular disease. The risk of recurrence of ischemic stroke was reported to be about 4 times higher in patients with a poor metabolizer or intermediate metabolizer genotype of the Cytochrome P450 2C19 genotype compared to the extensive metabolizer genotype. This genotypes of Cytochrome P450 2C19 were also different according to race.

The researches about cytochrome P450 2C19 genotype and clopidogrel resistance have been conducted mainly in patients with coronary artery disease and are not known in stroke patients. Few studies have examined whether the resistance of clopidogrel according to the genotype of cytochrome P450 2C19 in stroke patients is related to the occurrence and/or recurrence of cardiovascular disease. The hypothesis of this study is that "the poor metabolizer or intermediate metabolizer of the cytochrome P450 2C19 genotype in patients with acute ischemic stroke is associated with increased risk of cardiovascular disease and mortality compared to those who of extensive metabolizer of the cytochrome P450 2C19 genotype".

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic stroke confirmed by brain CT or MRI
2. Patient who received clopidogrel within 72 hours after onset of ischemic stroke
3. Adults over 19 years
4. Patients who agreed to participate in this study within 7 days after ischemic stroke
5. Patients who underwent Cytochrome P450 2C19 genotype test.

Exclusion Criteria:

1. Patients who currently take anticoagulation or is expected to take anticoagulation with 6 months from the screening date
2. Patients who need other antiplatelet drugs except aspirin and clopidogrel
3. Patients who were taking clopidogrel prior to ischemic stroke
4. Patients scheduled for coronary artery stenting, coronary artery bypass surgery, carotid endarterectomy, carotid and cerebral artery stenting
5. Patients with severe comorbidities or active cancer with an estimated life expectancy of less than two years
6. Patients who participated in other drug clinical trials within the past 30 days
7. Patients with high risk source of potential cardiac source of embolism in TOAST classification
8. Patients who are expected to unable to participate or continue the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ischemic stroke who received clopidogrel 75 mg to 300 mg (in the case of loading dose) within 24 hours of symptom onset and who underwent Cytochrome P450 2C19 genotyping test
Sampling Method: Non-Probability Sample
Enrollment: 2927 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
composite cardiovascular events | up to 6 months
  Occurrence of composite cardiovascular events (recurrent stroke, myocardial infarction, cardiovascular death)

SECONDARY OUTCOMES:
cardiovascular events | up to 6 months
  Occurrence of ischemic stroke
cardiovascular events | up to 6 months
  Occurrence of transient ischemic attack
cardiovascular events | up to 6 months
  Revascularization of cerebral, coronary, peripheral artery or aorta
cardiovascular events | up to 6 months
  Occurrence of myocardial infarction
early neurological worsening | up to 7 days
  increased National Institutes of Health Stroke Scale within 7 day after admission)
Prognosis | 3 months
  ratio of modified Rankin scale (0 - 2) at 3 months

OTHER OUTCOMES:
Incidence of major adverse events | Tile frame: participants will be followed at 0, 1, 3, 6 months
  Occurrence of major bleeding (fatal bleeding, symptomatic cerebral hemorrhage, ocular hemorrhage, bleeding which needs absolute bed rest or hospitalization or transfusion (more than 2 pack of whole blood or RBC).
  Occurrence of all-causes mortality

CONTACTS AND LOCATIONS:
Overall Officials: KyungYul Lee, Principal Investigator — Gangnam Severance Hospital
Locations (37):
- South Korea (37):
  - Yongin Severance Hospital, Yongin-si, Gyeonggi-do
  - Department of Neurology Korea University Ansan Hospital, Ansan
  - Department of Neurology Hallym University Sacred Heart Hospital, Anyang
  - Department of Neurology Inje University Busan Paik Hospital, Busan
  - Department of Neurology Dong-A University Hospital, Busan
  - Department of Neurology Kosin University Gospel Hospital, Busan
  - Department of Neurology Changwon Fatima Hospital, Changwon
  - Department of Neurology Hallym University Chuncheon Sacred Heart Hospital, Chuncheon
  - Department of Neurology Kangwon National University Hospital, Chuncheon
  - Department of Neurology Keimyung University Dongsan Hospital, Daegu
  - Department of Neurology Kyungpook National University Hospital, Daegu
  - Department of Neurology Daejeon Eulji Medical Center Eulji University, Daejeon
  - Department of Neurology Gimpo Woori Hospital, Gimpo-si
  - Department of Neurology National Health Insurance Service Ilsan Hospital, Goyang
  - Department of Neurology Myongji Hospital, Goyang
  - Department of Neurology Chosun University Hospital, Gwangju
  - Department of Neurology Chonnam National University Hospital, Gwangju
  - Department of Neurology Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si
  - Department of Neurology Wonkwang University Hospital, Iksan
  - Department of Neurology Gachon University Gil Medical Center, Incheon
  - Department of Neurology Inha University Hospital, Incheon
  - Department of Neurology Catholic Kwandong University International St.Mary's Hospital, Incheon
  - Department of Neurology Seoul National University Bundang Hospital, Seongnam
  - Department of Neurology Inje University Sanggye Paik Hospital, Seoul
  - Department of Neurology Seoul Medical Center, Seoul
  - Department of Neurology KyungHee University Hospital, Seoul
  - Department of Neurology Korea University Anam Hospital, Seoul
  - Department of Neurology Seoul National University Hospital, Seoul
  - Department of Neurology Severance Hospital, Yonsei University College of Medicine, Seoul
  - Department of Neurology National Medical Center, Seoul
  - Department of Neurology Hanyang University Seoul Hospital, Seoul
  - Department of Neurology KyungHee University Hospital at Gangdong, Seoul
  - Department of Neurology Kangdong Sacred Heart Hospital, Seoul
  - Department of Neurology, Gangnam Severance Hospital, Yonsei Univ. College of Medicine, Seoul
  - Department of Neurology Chung-Ang University Hospital, Seoul
  - Department of Neurology Ewha Womans University Seoul Hospital, Seoul
  - Department of Neurology Korea University Guro Hospital, Seoul

REFERENCES:
- [Background] Mitsios JV, Papathanasiou AI, Rodis FI, Elisaf M, Goudevenos JA, Tselepis AD. Atorvastatin does not affect the antiplatelet potency of clopidogrel when it is administered concomitantly for 5 weeks in patients with acute coronary syndromes. Circulation. 2004 Mar 23;109(11):1335-8. doi: 10.1161/01.CIR.0000124581.18191.15. Epub 2004 Mar 15. PMID 15023882
- [Background] Lau WC, Waskell LA, Watkins PB, Neer CJ, Horowitz K, Hopp AS, Tait AR, Carville DG, Guyer KE, Bates ER. Atorvastatin reduces the ability of clopidogrel to inhibit platelet aggregation: a new drug-drug interaction. Circulation. 2003 Jan 7;107(1):32-7. doi: 10.1161/01.cir.0000047060.60595.cc. PMID 12515739
- [Background] Nguyen TA, Diodati JG, Pharand C. Resistance to clopidogrel: a review of the evidence. J Am Coll Cardiol. 2005 Apr 19;45(8):1157-64. doi: 10.1016/j.jacc.2005.01.034. PMID 15837243
- [Background] Mega JL, Close SL, Wiviott SD, Shen L, Hockett RD, Brandt JT, Walker JR, Antman EM, Macias W, Braunwald E, Sabatine MS. Cytochrome p-450 polymorphisms and response to clopidogrel. N Engl J Med. 2009 Jan 22;360(4):354-62. doi: 10.1056/NEJMoa0809171. Epub 2008 Dec 22. PMID 19106084
- [Background] Simon T, Verstuyft C, Mary-Krause M, Quteineh L, Drouet E, Meneveau N, Steg PG, Ferrieres J, Danchin N, Becquemont L; French Registry of Acute ST-Elevation and Non-ST-Elevation Myocardial Infarction (FAST-MI) Investigators. Genetic determinants of response to clopidogrel and cardiovascular events. N Engl J Med. 2009 Jan 22;360(4):363-75. doi: 10.1056/NEJMoa0808227. Epub 2008 Dec 22. PMID 19106083
- [Background] Collet JP, Hulot JS, Pena A, Villard E, Esteve JB, Silvain J, Payot L, Brugier D, Cayla G, Beygui F, Bensimon G, Funck-Brentano C, Montalescot G. Cytochrome P450 2C19 polymorphism in young patients treated with clopidogrel after myocardial infarction: a cohort study. Lancet. 2009 Jan 24;373(9660):309-17. doi: 10.1016/S0140-6736(08)61845-0. Epub 2008 Dec 26. PMID 19108880
- [Background] Shuldiner AR, O'Connell JR, Bliden KP, Gandhi A, Ryan K, Horenstein RB, Damcott CM, Pakyz R, Tantry US, Gibson Q, Pollin TI, Post W, Parsa A, Mitchell BD, Faraday N, Herzog W, Gurbel PA. Association of cytochrome P450 2C19 genotype with the antiplatelet effect and clinical efficacy of clopidogrel therapy. JAMA. 2009 Aug 26;302(8):849-57. doi: 10.1001/jama.2009.1232. PMID 19706858
- [Background] Pan Y, Chen W, Xu Y, Yi X, Han Y, Yang Q, Li X, Huang L, Johnston SC, Zhao X, Liu L, Zhang Q, Wang G, Wang Y, Wang Y. Genetic Polymorphisms and Clopidogrel Efficacy for Acute Ischemic Stroke or Transient Ischemic Attack: A Systematic Review and Meta-Analysis. Circulation. 2017 Jan 3;135(1):21-33. doi: 10.1161/CIRCULATIONAHA.116.024913. Epub 2016 Nov 2. PMID 27806998
- [Background] Han SW, Kim YJ, Ahn SH, Seo WK, Yu S, Oh SH, Nam HS, Choi HY, Yoon SS, Kim SH, Lee JY, Lee JH, Hwang YH, Lee KO, Jung YH, Lee J, Sohn SI, Kim YN, Lee KA, Bushnell CD, Lee KY. Effects of Triflusal and Clopidogrel on the Secondary Prevention of Stroke Based on Cytochrome P450 2C19 Genotyping. J Stroke. 2017 Sep;19(3):356-364. doi: 10.5853/jos.2017.01249. Epub 2017 Sep 29. PMID 29037010
- [Background] Lee SS, Lee SJ, Gwak J, Jung HJ, Thi-Le H, Song IS, Kim EY, Shin JG. Comparisons of CYP2C19 genetic polymorphisms between Korean and Vietnamese populations. Ther Drug Monit. 2007 Aug;29(4):455-9. doi: 10.1097/FTD.0b013e31811f383c. PMID 17667801
- [Background] Wang Y, Zhao X, Lin J, Li H, Johnston SC, Lin Y, Pan Y, Liu L, Wang D, Wang C, Meng X, Xu J, Wang Y; CHANCE investigators. Association Between CYP2C19 Loss-of-Function Allele Status and Efficacy of Clopidogrel for Risk Reduction Among Patients With Minor Stroke or Transient Ischemic Attack. JAMA. 2016 Jul 5;316(1):70-8. doi: 10.1001/jama.2016.8662. PMID 27348249
- [Background] CAPRIE Steering Committee. A randomised, blinded, trial of clopidogrel versus aspirin in patients at risk of ischaemic events (CAPRIE). CAPRIE Steering Committee. Lancet. 1996 Nov 16;348(9038):1329-39. doi: 10.1016/s0140-6736(96)09457-3. PMID 8918275
- [Derived] Jung YH, Song TJ, Kim J, Park HK, Han SW, Kim YD, Park JH, Cha JK, Park HY, Sohn SI, Yu S, Lee JH, Shin DH, Kim EG, Lee HS, Lee KY; PLATELET Trial Investigators. Cytochrome P450 2C19 Genotypes and Clopidogrel in Patients With Ischemic Stroke: A Nonrandomized Clinical Trial. JAMA Netw Open. 2025 Apr 1;8(4):e250398. doi: 10.1001/jamanetworkopen.2025.0398. PMID 40184070
- [Derived] Song TJ, Kim J, Han SW, Kim YD, Lee JY, Ahn SH, Lee HS, Jung YH, Lee KY. Clopidogrel preventive effect based on cytochrome P450 2C19 genotype in ischaemic stroke: protocol for multicentre observational study. BMJ Open. 2020 Aug 5;10(8):e038031. doi: 10.1136/bmjopen-2020-038031. PMID 32759249